CLINICAL TRIAL: NCT03053011
Title: Alarm Relay Bracelet for Simplification and Security Respiratory Assistance at Home: Evaluation of the Nocturnal Awakening Capability in Ventilated Patients and Healthy Volunteers
Brief Title: Evaluation of the Awakening Capability by a Vibrating Bracelet (BRASSARD)
Acronym: BRASSARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association Nationale pour les Traitements A Domicile, les Innovations et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-A01044-47
Record Dates: First submitted 2017-02-02; First posted 2017-02-14 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Congenital Central Hypoventilation Syndrome; Patients With Nocturnal Ventilatory Assistance; Healthy Volunteers
MeSH Terms: conditions — Congenital central hypoventilation syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vibrating bracelet (Experimental): A bracelet with vibrations triggered randomly overnight
  Interventions: Other: Vibrating bracelet

INTERVENTIONS:
Other: Vibrating bracelet — A bracelet with vibrations triggered randomly overnight. The sleeper's awakening capability will be evaluated each time the bracelet vibrates (5 times in the night).

SUMMARY:
As part of developing a relay alarm project, the aim of the study is to test a sleeper's capability to wake up via a vibrating alarm around the wrist (vibrating bracelet).

ELIGIBILITY:
Inclusion Criteria:

* speak french
* with social security For healthy volunteers : no sleep disorder, known neurological or respiratory pathology For patients : congenital central hypoventilation syndrome or ventilatory assistance whatever the indication, able to act on their ventilator, and in stable state on the respiratory level for at least 3 months.

Exclusion Criteria:

* subjects taking treatment that may interfere with sleep patterns
* intake of alcohol or any substance (alcohol, drugs) that may interfere with sleep patterns the day before the polysomnography

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
Total awakening capability | 1 night
  Proportion of the activations of the bracelet causing an awakening sufficient for the subject to stop the application and do a cognitive task : note the wake-up time

SECONDARY OUTCOMES:
Awakening capability in each stage of sleep | 1 night
  Proportion of awakenings in different stages of sleep (slow wave sleep, Rapid Eye Movement sleep) relative to the total number of vibrations triggering by the bracelet
Awakening without capability to do the cognitive task | 1 night
  Proportion of the activations of the bracelet causing an awakening without the cognitive task

CONTACTS AND LOCATIONS:
Overall Officials: Valérie ATTALI, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service des pathologies du sommeil - GH Pitié-Salpêtrière, Paris, France